CLINICAL TRIAL: NCT04991662
Title: Effect of Three Weight-adjusted Vasopressors for With Combined Spinal-Epidural Anesthesia for Elective Cesarean Delivery: A Randomized Controlled Trial
Brief Title: Effect of Three Weight-adjusted Vasopressors for Elective Cesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Chao Xu, Head of Otolaryngology, Xuzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SFY2021-HZ08-11
Record Dates: First submitted 2021-06-09; First posted 2021-08-05 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-09

CONDITIONS: Cesarean Section Complications
MeSH Terms: interventions — Metaraminol; Phenylephrine; Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- metaraminol group (Experimental): During the cesarean section, metaraminol 2ug/kg/min is preventively infused after anesthesia to prevent and treat hypotension.
  Interventions: Drug: metaraminol
- phenylephrine group (Experimental): During cesarean section, preventive infusion of phenylephrine 0.54ug/kg/min after anesthesia to prevent and treat hypotension.
  Interventions: Drug: Phenylephrine
- norepinephrine group (Experimental): During cesarean section, preventive infusion of norepinephrine 0.08ug/kg/min after anesthesia to prevent and treat hypotension.
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: metaraminol — Infusion of metaraminol adjusted according to body weight to obtain higher pH value of fetal umbilical artery blood.
  Other Names: M group
  Arms: metaraminol group
Drug: Phenylephrine — Infusion of Phenylephrine adjusted according to body weight to obtain higher pH value of fetal umbilical artery blood.
  Other Names: P group
  Arms: phenylephrine group
Drug: Norepinephrine — Infusion of Norepinephrine adjusted according to body weight to obtain higher pH value of fetal umbilical artery blood.
  Other Names: N group
  Arms: norepinephrine group

SUMMARY:
This study compared the effects of prophylactic infusion of metaraminol, phenylephrine and norepinephrine adjusted according to body weight on fetal acid-base balance and maternal hemodynamics.

DETAILED DESCRIPTION:
At present, the ED90 of metaraminol, phenylephrine, and norepinephrine in the prevention of cesarean section hypotension has been explored. We compare the effects of three drugs on the fetus and mothers at the concentration of ED90 to provide advice on the use of vasoactive drugs for obstetrics anesthesia .

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnancy at term scheduled to be delivered via elective cesarean delivery;
2. height 150-180 cm;
3. American Society of Anesthesiologists (ASA) physical status II-III;
4. body mass index (BMI) <35 kg/m2.

Exclusion Criteria:

1. transverse presentation, fetal macrosomia;
2. uterine abnormalities (eg, large fibroids, bicornuate uterus);
3. polyhydramnios;
4. ruptured membranes, oligohydramnios;
5. intrauterine growth restriction;
6. gestational or nongestational hypertension, diabetes, or eclampsia;
7. hypertensive disorders or any condition associated with autonomic neuropathy (such as diabetes mellitus for >10 years) or renal failure;
8. contraindications for combined spinal-epidural anesthesia;
9. participants who declined to sign informed consent forms.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Umbilical artery blood pH | 30 seconds after delivery
  pH value of fetal umbilical artery blood

SECONDARY OUTCOMES:
hypotension | Intraoperative
  Number of Participants with systolic blood pressure reduction >20% baseline value or systolic blood pressure <90 mm Hg before delivery
bradycardia | Intraoperative
  Number of Participants with heart rate was ≤50 bpm before delivery
The incidence of nausea in pregnant women | Intraoperative
  Anesthesiologist observes combined patient dictation.
Umbilical artery blood base excess | 30sec after delivery
  base excess of fetal umbilical artery blood
The incidence of vomiting in pregnant women | Intraoperative
  Anesthesiologist observes combined patient dictation

CONTACTS AND LOCATIONS:
Overall Officials: Feng Yi, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Department of Anesthesiology and Operating Room, Affiliated Hospital of Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No